CLINICAL TRIAL: NCT07006415
Title: Brain-computer Interface Rehabilitation And Virtual Environments in Functional Neurological Disorder (BRAVE-FND)
Acronym: BRAVE-FND
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 349392; TBC (Other Grant/Funding Number: TBC)
Record Dates: First submitted 2025-05-19; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Functional Neurological Disorder; Conversion Disorder; Functional Neurological Disorders; Conversion Disorder With Weakness/Paralysis
Keywords: brain-computer interface; rehabilitation
MeSH Terms: conditions — Conversion Disorder; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain-computer interface rehabilitation (Experimental): Brain-computer interface rehabilitation
  Interventions: Device: Brain-computer interface rehabilitation

INTERVENTIONS:
Device: Brain-computer interface rehabilitation — 10 sessions of motor imagery rehearsal rehabilitation using a brain-computer interface with functional electrical stimulation and a virtual avatar

SUMMARY:
The purpose of this study is to determine whether a course of rehabilitation using a device called a brain-computer interface can change the level of control people feel over bodily movements, in functional neurological disorder.

ELIGIBILITY:
Inclusion Criteria:

* DSM5 diagnosis of motor FND (limb weakness, gait disorder, tremor or dystonia) from a neurologist and/or neuropsychiatrist.
* Moderate or severe symptoms (≥4 on Clinical Global Impression Severity (CGI-S) scale).
* Able to tolerate VR and BCI use.
* Age 18 - 60 years.
* English speaking.

Exclusion Criteria:

* Current diagnosis of epilepsy, severe depression, bipolar disorder, psychotic disorder, personality disorder, or drug/alcohol dependence/harmful use (defined as meeting DSM-5 criteria) (Mini International Neuropsychiatric Interview [MINI] 7.0). Positive diagnoses on the MINI will be subject to confirmation at clinical interview by a psychiatrist.
* Current diagnosis of epilepsy, autistic spectrum disorder, dementia, learning disability (defined as meeting DSM-5 criteria) based on clinical interview by a psychiatrist.
* A pacemaker, implantable cardioverter-defibrillator or any other implanted electronic or metallic device.
* Current pregnancy.
* Non-registration with a GP or failure to consent to sharing of the GP summary care record and any psychiatric assessments held.
* Those enrolled in another clinical or research study.
* Those unable to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in sense of agency over limb movements | Baseline (same day as rehabilitation session 1, immediately before session) and after course of 10 sessions of brain-computer interface rehabilitation (same day as rehabilitation session 10, immediately after session) (intra-subject)
  Seven point Likert scale for explicit self-reported sense of agency over limb movements